CLINICAL TRIAL: NCT02199067
Title: Measurement of Exhaled Propofol During a Total Intravenous Anesthesia With Propofol and Remifentanil
Brief Title: Measurement of Exhaled Propofol
Acronym: PIAG1
Status: Terminated | Type: Observational
Why Stopped: technical difficulties of probe measurement
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Tino Münster, Prof. Dr., University of Erlangen-Nürnberg Medical School
Other Study IDs: PIAG1
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Anaesthesia With Propofol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — arterial blood samples (serum)
Oversight: Data Monitoring Committee: No

SUMMARY:
Propofol is a common intravenous anaesthetic drug used for anaesthesia induction and for permanent infusion to maintain anaesthesia (total intravenous anaesthesia). Different to the volatile anaesthetics (feedback concentrations in exhaled breathing gas) piloting of an total intravenous anaesthesia with propofol is done only by experience of the anaesthetist or according to pharmacokinetic models. In this study we want to investigate if the exhaled fraction of propofol is a potential measurement parameter for piloting anaesthesia. Exhaled propofol will be measured with an electrochemical sensor developed by "Drägerwerk AG & Co. KGaA". Exhaled propofol levels will be compared with the corresponding arterial serum concentrations of propofol. Furthermore we investigate the correlation of exhaled propofol levels with the Bispectral Index (BIS).

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anaesthesiologists) classification I & II
* Body-Mass-Index < 35
* elective surgery with the necessity of an arterial catheter

Exclusion Criteria:

* chronic obstructive lung disease
* bronchial asthma
* smokers with more than 5 packyears
* peripheral artery occlusive disease
* diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patients undergoing elective surgery
  * total intravenous anaesthesia
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
exhaled propofol levels in breathing gas | continous recording during the whole anaesthesia (duration depents on surgery, between 2 and 12 hours)

SECONDARY OUTCOMES:
propofol concentration in arterial blood serum | samples taken during anaesthesia (13 blood samples), duration of anaesthesia depends on surgery, 2 to 12 hours
Bispectral Index (BIS) | continous recording during the whole anaesthesia (duration depents on surgery, between 2 and 12 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Schmidt S, Ihmsen H, Munster T, Schuttler J, Jeleazcov C, Wehrfritz A. Determination of the Long-Term Stability of Propofol in Human Plasma Frozen for Eight Years and Quantified by UHPLC-MS/MS. Int J Anal Chem. 2025 Aug 22;2025:7533068. doi: 10.1155/ianc/7533068. eCollection 2025. PMID 40895257